CLINICAL TRIAL: NCT05465122
Title: Long-Term Observational Extension of Participants in the CREST-2 Randomized Clinical Trial
Brief Title: CREST-2 Long-term Observational Extension Study
Acronym: C2LOE
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Alabama at Birmingham (Other); University of Maryland (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, James F. Meschia, Principal Investigator, Mayo Clinic
Other Study IDs: 21-007363; 1U01NS119169-01A1 (NIH)
Record Dates: First submitted 2022-06-30; First posted 2022-07-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Stenoses, Carotid
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Carotid Stenting Group (CAS): Subjects assigned to the intensive medical management with carotid stenting group in the CREST-2 study (NCT02089217)
  Interventions: Procedure: FDA-approved carotid stents; Other: Intensive Medical Management
- Carotid Endarterectomy Group (CEA): Subjects assigned to the intensive medical management with carotid endarterectomy group in the CREST-2 study (NCT02089217)
  Interventions: Procedure: Carotid Endarterectomy; Other: Intensive Medical Management
- Intensive Medical Management Group - no CAS: Subjects assigned to the intensive medical management alone with no carotid stenting (CAS) group in the CREST-2 study (NCT02089217)
  Interventions: Other: Intensive Medical Management
- Intensive Medical Management Group - no CEA: Subjects assigned to the intensive medical management alone with no carotid endarterectomy (CEA) group in the CREST-2 study (NCT02089217)
  Interventions: Other: Intensive Medical Management

INTERVENTIONS:
Procedure: Carotid Endarterectomy — This is the standard proven therapy for carotid stenosis that involves an arteriotomy followed by removal of plaque and reconstruction of the vessel.
  Groups: Carotid Endarterectomy Group (CEA)
Procedure: FDA-approved carotid stents — This is the standard proven therapy for carotid stenosis that involves an arteriotomy followed by removal of plaque and reconstruction of the vessel.
  Groups: Carotid Stenting Group (CAS)
Other: Intensive Medical Management — INTERVENT risk factor management program to help manage patient's risk factors. The INTERVENT program will provide individualized risk factor counseling sessions (via telephone or internet) at regular interval by healthcare workers who are specially trained to help patients follow the medical management plan.

SUMMARY:
The purpose of this Long-Term Observational Extension of Participants in the CREST-2 Randomized Clinical Trial (C2LOE - ClinicalTrials.gov Identifier: NCT02089217) study is to study is to assess post-procedural efficacy of carotid endarterectomy and carotid stenting.

DETAILED DESCRIPTION:
Atherosclerotic plaque in the carotid arteries is responsible for 10 to 15% of all ischemic strokes. The ongoing NINDS-funded CREST-2 multicenter randomized clinical trial is testing whether in the short term (up to 4 years after study entry) procedural revascularization improves stroke prevention above and beyond what can be achieved with intensive medical management of vascular risk factors, especially hypertension and hyperlipidemia. Our proposal is for an observational extension of the CREST-2 clinical trial to test whether revascularization improves stroke prevention in the clinically relevant long term (up to 8 to 10 years). The current application proposes to use a site-less, centralized telephone approach to extend the follow-up of CREST-2 trial participants for assessing the primary study outcome (stroke) for up to 10 years. The average follow-up will increase from between 2-3 years (clinic-based randomized trial) to 7-8 years (observational extension). Each patient will be contacted by telephone at 6-month intervals, and queried regarding all hospitalizations since the last contact. Suspected stroke events will be adjudicated by an expert clinical events committee based on medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Currently active or graduated participants in the CREST-2 randomized trial
* Able to provide written informed consent by self
* Fluent in English or Spanish

Exclusion Criteria:

* Unable to provide written informed consent
* Inability to follow study procedures

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with asymptomatic carotid stenosis previously randomized in the CREST-2 trial.
Sampling Method: Non-Probability Sample
Enrollment: 2480 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Stroke | 5 years
  Number of participants to experience a stroke

CONTACTS AND LOCATIONS:
Overall Officials: James Meschia, MD, Principal Investigator — Mayo Clinic
Locations (64):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Pheonix, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Central Arkansas VA, Little Rock, Arkansas
  - Mission Cardiovascular Research Institute, Fremont, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - USC/Keck Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Kaiser Permanente Divsion of Research, San Francisco, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - St. Joseph's Medical Center, Stockton, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Morton Plant Mease Healthcare, Clearwater, Florida
  - University of Florida Health at Shands, Gainesville, Florida
  - Lyerly Neurosurgery/Baptist Health, Jacksonville, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Miami Cardiac and Vascular Institute, Miami, Florida
  - Cardiovascular Institute NW Florida, Panama City, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Endeavor Health/NorthShore University, Evanston, Illinois
  - Prairie Heart/St. John's Hospital, Springfield, Illinois
  - Deaconess Heart Group, Newburgh, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Baptist Health, Lexington, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - VA Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - White Oak Medical Center, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - VA Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan Vascular Center, Flint, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - North Memorial Medical Center, Golden Valley, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mercy Hospital, St Louis, Missouri
  - SUNY Buffalo, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Crouse Hospital, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Mercy Health St. Vincent, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - VA Pittsburgh, Pittsburgh, Pennsylvania
  - Berks Cardiologists, Wyomissing, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Tennova Healthcare, Knoxville, Tennessee
  - Seton Medical Center, Austin, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - VA Puget Sound, Seattle, Washington
  - Gundersen Clinic, Ltd., La Crosse, Wisconsin
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials